CLINICAL TRIAL: NCT03677323
Title: Evaluation of the Efficacy of VR on Pain and Anxiety When Performing an Ultrasound-controlled Ankle Block.
Acronym: VRBLOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Jean, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL2017-TP02
Record Dates: First submitted 2018-09-13; First posted 2018-09-19 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Hallux Valgus; Surgery
Keywords: virtual reality; pain; anxiety
MeSH Terms: conditions — Hallux Valgus; Pain; Anxiety Disorders | interventions — Droperidol; Propofol; Sufentanil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): The virtual reality device will consist of the virtual reality headset and headphones for full immersion.
  Interventions: Device: Virtual reality
- Drug sedation (Active Comparator): The sedation group will benefit from drug sedation used in current practice, that is to say an association of Sufentanil, Droleptan and Propofol.
  Interventions: Drug: Droleptan; Drug: Propofol; Drug: Sufentanyl

INTERVENTIONS:
Device: Virtual reality — The patient will have the choice between different environments and the use of this device will remain under the control of the medical team.
  The patient will wear the virtual reality device at the time of the completion of the ankle block and will remove it once the nerve puncture is complete.
  Other Names: VR
  Arms: Virtual reality
Drug: Droleptan — Venous administration of 1.25 mg of Droleptan
  Other Names: Sedation
  Arms: Drug sedation
Drug: Propofol — Venous administration of 20 mg of Propofol
  Other Names: Sedation
  Arms: Drug sedation
Drug: Sufentanyl — Venous administration of 5 μg of Sufentanyl.
  Other Names: Sedation
  Arms: Drug sedation

SUMMARY:
The purpose of this study is to observe or not a reduction on pain and anxiety felt by the patient when performing an ultrasound-controlled ankle block in preparation for forefoot surgery, using a virtual reality device instead of drug sedation.

DETAILED DESCRIPTION:
Currently, in preparation for forefoot surgery, the realization of the ankle block is accompanied by drug sedation.

The investigator's randomized study aims to compare the anxiety and pain experienced by patients who have benefited from drug sedation with those of patients who benefited from the virtual reality device at the time of the realization of the ankle block.

ELIGIBILITY:
Inclusion Criteria:

* Patient with medical insurance
* Major patient requiring a Hallux Valgus surgery
* Patient who received information about study and signes a consent to participate in the study

Exclusion Criteria:

* Minor patient
* Patient participating in another interventional study
* Patient refusing to sign the consent form
* Patient for whom it is impossible to give informed information
* Patient who had previously undergone forefoot surgery under locoregional anesthesia
* Patient with poor skin condition or infection at puncture sites
* Patient refusing locoregional anesthesia
* Patient under the protection of justice, under curatorship or under tutorship
* Patient undergoing anxiolytic or antidepressant treatment
* Photosensitive epileptic patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Digital visual scale to assess pain of patients during the treatment | 5 min after the first nerve punction
  Numeric scale numbered from 0 to 10. 0: no pain 10 : worst possible pain
Digital visual scale to assess anxiety of patients during the treatment | 5 min after the first nerve punction
  Numeric scale numbered from 0 to 10. 0: no anxiety 10 : worst possible anxiety

SECONDARY OUTCOMES:
Patient satisfaction questionnaire | 5 min after the last nerve punction
  Concerns all patients Numeric scale numbered from 0 to 10. 0: unsatisfied 10 : very satisfied
Patient comfort assessment questionnaire | 5 min after the last nerve punction
  Concerns all patients. This is a question to determine their comfort levels during the experiment. Numeric scale numbered from 1 to 5.
  1. : very comfortable
  2. : comfortable
  3. : less comfortable
  4. : uncomfortable
  5. : very uncomfortable

CONTACTS AND LOCATIONS:
Overall Officials: Thomas PILLANT, MD, Principal Investigator — Clinique Saint Jean, Montpellier
Locations (1):
- Clinique Saint Jean, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mosso JL, Gorini A, De La Cerda G, Obrador T, Almazan A, Mosso D, Nieto JJ, Riva G. Virtual reality on mobile phones to reduce anxiety in outpatient surgery. Stud Health Technol Inform. 2009;142:195-200. PMID 19377147
- [Background] Furman E, Jasinevicius TR, Bissada NF, Victoroff KZ, Skillicorn R, Buchner M. Virtual reality distraction for pain control during periodontal scaling and root planing procedures. J Am Dent Assoc. 2009 Dec;140(12):1508-16. doi: 10.14219/jada.archive.2009.0102. PMID 19955069
- [Background] Patterson DR, Jensen MP, Wiechman SA, Sharar SR. Virtual reality hypnosis for pain associated with recovery from physical trauma. Int J Clin Exp Hypn. 2010 Jul;58(3):288-300. doi: 10.1080/00207141003760595. PMID 20509069
- [Background] Nilsson S, Finnstrom B, Kokinsky E, Enskar K. The use of Virtual Reality for needle-related procedural pain and distress in children and adolescents in a paediatric oncology unit. Eur J Oncol Nurs. 2009 Apr;13(2):102-9. doi: 10.1016/j.ejon.2009.01.003. Epub 2009 Feb 20. PMID 19230769
- [Background] Konstantatos AH, Angliss M, Costello V, Cleland H, Stafrace S. Predicting the effectiveness of virtual reality relaxation on pain and anxiety when added to PCA morphine in patients having burns dressings changes. Burns. 2009 Jun;35(4):491-9. doi: 10.1016/j.burns.2008.08.017. Epub 2008 Dec 27. PMID 19111995
- [Background] Wright JL, Hoffman HG, Sweet RM. Virtual reality as an adjunctive pain control during transurethral microwave thermotherapy. Urology. 2005 Dec;66(6):1320. doi: 10.1016/j.urology.2005.06.123. PMID 16360473
- [Background] Burt DE. Virtual reality in anaesthesia. Br J Anaesth. 1995 Oct;75(4):472-80. doi: 10.1093/bja/75.4.472. No abstract available. PMID 7488491